CLINICAL TRIAL: NCT06644014
Title: Guidance with Oura and AI for Reducing Arterial Stiffness - the GONDOR-AS Trial
Brief Title: Reducing Arterial Stiffness with a Smart Ring and AI-Guided Exercise
Acronym: GONDOR-AS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pauli Ohukainen (Industry)
Collaborators: Kuopio Research Institute of Exercise Medicine (Other)
Responsible Party: Sponsor-Investigator, Pauli Ohukainen, Senior Research Scientist, Ouraring Inc.
Organization: Ouraring Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 207/13.00/2024
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Arterial Stiffness; Maximal Oxygen Uptake
Keywords: arterial stiffness; maximal oxygen uptake; HIIT training; Oura Ring; Oura; AI; Artificial Intelligence; Aerobic Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Note: Participants are blinded to the outcome measure (CVA) on their Oura App. Outcomes are analyzed by blinded researchers not actively involved in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AI-instructed group (Experimental): Participants in this group will receive Oura Rings and access to AI-based exercise guidance. They are instructed to follow received instructions, but they are blinded to their outcome measure (CVA).
  Interventions: Behavioral: Exercise
- Supervised exercise group (Active Comparator): Participants in this group receive Oura Rings and are instructed to attend supervised HIIT-cycling sessions twice a week. They are blinded to their outcome measure (CVA).
  Interventions: Behavioral: Exercise
- Ring-only group (Other): Participants in this group receive Oura Rings but no AI-advice or supervised training. They are blinded to the outcome measure (CVA).
  Interventions: Device: Smart Ring

INTERVENTIONS:
Behavioral: Exercise — Participant will communicate with a "chatbot-like" proprietary AI to receive exercise instructions. The AI will provide personalized advice according to the user's needs, aiming for 2-3 hours of steady-state zone 2 -effort aerobic exercise. Instructions will also be tailored to the user's exercise preferences and limitations (for example, suggest cycling, if running is not convenient).
  Arms: AI-instructed group
Behavioral: Exercise — Supervised HIIT -cycling twice a week. Intensities for cycling intervals will are based on the participants fitness-level determined at first visit. Intensity will gradually increase over the 12-week period
  Arms: Supervised exercise group
Device: Smart Ring — Participants will only receive an Oura Ring, but will not change anything about their normal physical activity.
  Arms: Ring-only group

SUMMARY:
The goal of this three-month clinical trial is to study if wearing an Oura Ring and following the exercise guidance provided by an AI-based Advisor in the Oura App works to reduce arterial stiffness. It will also study the difference between different exercise protocols in reducing arterial stiffness and improving aerobic fitness. The main questions the study aims to answer are:

* Can an AI-based Advisor provide useful exercise guidance that helps improve cardiovascular health and aerobic fitness?
* Does regular exercise lower arterial stiffness measured with a clinical reference device and Oura Ring's proprietary Cardiovascular Age -metric and its estimated arterial stiffness?
* Is there a difference between attending supervised high-intensity interval (HIIT) training sessions and following personalized exercise instructions for steady-state aerobic training?

Participants will:

* Follow Oura's AI Advisor's instructions at their own convenience, attend supervised training sessions, or just wear the Ring without changing their lifestyle
* Visit an exercise physiology lab in the beginning of the trial and after three months for measurements in arterial stiffness, cardiorespiratory fitness, and body composition

In addition, the study contains questionnaires investigating the participants' experiences related to lifestyle changes.

DETAILED DESCRIPTION:
This is a single-site, 12-week randomized, controlled trial (RCT) consisting of three groups (N = 55 per group):

* The Oura Ring (a control group)
* The Oura Ring + Supervised high-intensity interval training (HIIT) twice a week
* The Oura Ring + AI-based Coaching for steady-state aerobic training (no external supervision)

Exercise modalities are selected based on hypothesized long-term sustainability and expected cardiorespiratory outcomes. The HIIT protocol has been tested in previous studies and found to be effective in improving VO2max; but it is unlikely to be sustainable in the long-term. Thus, in this study we compare the HIIT protocol to individualized, steady-state ("Zone 2") exercise guidance provided by AI.

Participants will be recruited via e-mail and newspaper ads from the region of Kuopio, Finland. All groups will be blinded to their CVA/PWV information but will use identical Rings. Apart from the AI coach -group, Oura Ring App experiences will also be identical. The study consists of four (4) visits.

The study site is Kuopio Institute for Exercise Medicine, Kuopio, Finland. Participants will be provided materials for an informed consent prior to participation. Eligible participants who have provided a written consent will be invited for the first baseline measurement (Visit 1) where they will be provided Oura Rings and given instructions for using it, and their VO2max is measured. The next baseline measurement (Visit 2) is scheduled for two weeks which is the time the Ring needs to calibrate its Cardiovascular Age and pulse-wave velocity (PWV) estimates. At the second baseline measurement, the participants' PWV is recorded with a reference device and their body composition is also measured. Following these measurements, they are immediately randomized to one of the three study groups and given written and oral instructions specific to their allocation. After 12 weeks, the participant is invited for a repeated VO2max measurement (Visit 3), followed by final PWV and body composition measurements (Visit 4) within the same week. Measurements are not conducted on the same days due to fasting requirements for PWV, and interfering effect of VO2max testing on PWV.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported moderate intensity physical activity less than 2 hours 30 minutes per week or vigorous intensity physical activity less than 1 hour 15 minutes per week.

Exclusion Criteria:

* Coronary artery disease (or other chronic condition preventing safe participation in an exercise intervention), diabetes and moderate/severe hypertension diagnosed by a physician. Inability to use the Oura Ring for some reason (e.g. work-related restrictions) is also considered as exclusion criteria; however, short interruptions (e.g. 1-2 hour work tasks without ring) are possible.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness, clinical reference | Three months
  Measurement of carotid-femoral pulse-wave velocity (PWV) using the Complior device (Alam Medical)
VO2max | Three months
  Maximal oxygen consumption measured while cycling with an ergometer (Ergoselect 4, Ergoline GmbH, Germany), and VO2max will be measured by the breath-by-breath method (Vyntus CPX, Vyaire Medical, USA)

SECONDARY OUTCOMES:
Estimated PWV | Three months
  Estimation of PWV using Oura Ring's proprietary photophletysmogram -based algorithm
Change in Cardiovascular Age | Three months
  The delta (change) in Oura Ring's proprietary Cardiovascular Age metric, which is expressed as a difference between their chronological age and cardiovascular age (units are plus- and minus- age years; e.g. -3 years).

OTHER OUTCOMES:
Change in body weight | Three months
  Difference between baseline- and post-intervention weight (measured by Inbody 720 -device, South Korea)
Change in body fat | Three months
  Difference between baseline- and post-intervention body fat mass (measured by Inbody 720 -device, South Korea)
Change in muscle mass | Three months
  Difference between baseline- and post-intervention muscle mass (measured by Inbody 720 -device, South Korea)

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio Institute of Exercise Medicine, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan will be updated pending the Sponsor's (Ouraring ltd) finalization of the relevant data sharing standards and practices